CLINICAL TRIAL: NCT00006477
Title: Phase I Clinical Trial of Recombinant Viscumin (rVISCUMIN, rMISTLETOE LECTIN, rML) Administered Twice Weekly by the Subcutanous Route in Patients With Solid Tumors After Failure of Standard Therapy
Brief Title: Mistletoe Lectin in Treating Patients With Refractory Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-13001; EORTC-13001
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Dietary Supplement: mistletoe extract

SUMMARY:
RATIONALE: Mistletoe lectin may slow the growth of cancer cells and be an effective treatment for solid tumors.

PURPOSE: Phase I trial to study the effectiveness of mistletoe lectin in treating patients who have refractory advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of mistletoe lectin (recombinant viscumin) in patients with advanced solid tumors who have failed standard therapy.
* Determine the optimal biologically active dose of mistletoe lectin based on analysis of specific biological surrogate markers, including plasma cytokine levels and peripheral counts of activated immune cells and immunological stimulation at the RNA level of the immune cells.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine whether induction of antibodies against mistletoe lectin occurs in these patients.
* Determine whether modification of endothelial parameters occurs in patients treated with this regimen.
* Determine the objective response rates in patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive mistletoe lectin (recombinant viscumin) subcutaneously twice weekly. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of mistletoe lectin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Additional patients are treated at the highest dose level immediately preceding the MTD.

Patients are followed every 3 months until disease progression or initiation of another therapy.

PROJECTED ACCRUAL: A maximum of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven progressive advanced solid tumor that is not amenable to standard therapy (i.e., resistant to standard therapy or for which no standard therapy exists)
* No clinically symptomatic CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT less than 2 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase less than 2 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine less than 1.4 mg/dL

Cardiovascular:

* No ECG abnormalities of clinical relevance

Other:

* No severe or unstable systemic disease or infection
* No circumstances (e.g., alcoholism or substance abuse) that would preclude study
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunostimulating substances (e.g., biologic response modifiers or colony-stimulating factors)
* No concurrent immunostimulating substances (e.g., biologic response modifiers or colony-stimulating factors (except in life-threatening situations))

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* At least 4 weeks since prior systemic steroids
* At least 4 weeks since prior hormonal therapy
* No concurrent systemic steroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No prior mistletoe preparations
* At least 4 weeks since prior investigational treatment
* No other concurrent anticancer agents
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-09; Primary Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Aamdal, MD, PhD, Study Chair — Norwegian Radium Hospital
Locations (2):
- Klinikum der J.W. Goethe Universitaet, Frankfurt, Germany
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Bergmann L, Aamdal S, Marreaud S, Lacombe D, Herold M, Yamaguchi T, Wilhelm-Ogunbiyi K, Lentzen H, Zwierzina H; European Organisation for Research and Treatment of Cancer. Phase I trial of r viscumin (INN: aviscumine) given subcutaneously in patients with advanced cancer: a study of the European Organisation for Research and Treatment of Cancer (EORTC protocol number 13001). Eur J Cancer. 2008 Aug;44(12):1657-62. doi: 10.1016/j.ejca.2008.05.005. Epub 2008 Jul 2. PMID 18602257